CLINICAL TRIAL: NCT03683355
Title: Characterization of Radiolabeled Tracer Uptake Pattern in Noninfected Transcatheter Aortic Valves. The COUNT Study. A Prospective, Observational Study.
Brief Title: Characterization of RadiOlabeled Tracer Uptake Pattern in Noninfected Transcatheter Aortic Valves.
Acronym: COUNT
Status: Active, not recruiting | Type: Observational
Sponsor: Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec (Other)
Responsible Party: Principal Investigator, Josep Rodes-Cabau, Principal Investigator, Centre de Recherche de l'Institut Universitaire de Cardiologie et de Pneumologie de Quebec
Organization: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Other Study IDs: COUNT
Record Dates: First submitted 2018-09-11; First posted 2018-09-25 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Infective Endocarditis
Keywords: Transcatheter aortic valve replacement; Infective endocarditis; Radionuclide imaging; Radiolabeled tracer uptake pattern
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Edwards Sapien 3: Patients who underwent transcatheter aortic valve replacement with the Edwards Sapien 3 valve
  Interventions: Radiation: 18F-FDG PET/CT
- Core Valve Evolut R: Patients who underwent transcatheter aortic valve replacement with the Core Valve Evolut R valve
  Interventions: Radiation: 18F-FDG PET/CT

INTERVENTIONS:
Radiation: 18F-FDG PET/CT — 18F-FDG PET/CT and blood cultures will be performed at 3-month follow-up after TAVR Patients with positive 18F-FDG PET/CT (moderate or intense radiolabeled tracer uptake) will be scheduled for a second 18F-FDG PET/CT at 6-month follow-up.

SUMMARY:
Therefore, the objective of the study is to characterize the pattern of radiolabeled tracer (18F-FDG) uptake in noninfected transcatheter heart valves in early follow-up after transcatheter aortic valve replacement (TAVR).

DETAILED DESCRIPTION:
Diagnostic accuracy of Infective endocarditis (IE) is commonly challenging. Current clinical guidelines recommend the use of the modified Duke criteria, based on clinical, echocardiographic and biological findings, as well as the results of blood cultures and serologies. Advances in imaging techniques have resulted in an improvement in the identification of endocardial involvements and extracardiac complications of IE. Thus, recent works have demonstrated that 18F-FDG PET/CT and radiolabeled leucocyte SPECT/CT may improve the detection of silent endocardial lesions. The sites of radiotracer accumulation show regions of a high metabolic activity due to an inflammation or infection process. It is well known that, in surgical prosthetic valves, a mild radiotracer uptake in the perivalvular area may occur in the absence of infection and could therefore be considered as a normal pattern, particularly early after valve replacement. However, evidence of this phenomenon is lacking regarding transcatheter heart valves and the factors used to distinguish between normal and abnormal patterns of radiolabeled tracer are not standardized. The hypothesis is that patients undergoing transcatheter aortic valve replacement (TAVR) show a radiolabeled tracer (18F-FDG) uptake around the prosthesis despite the absence of IE. Moreover, the uptake pattern might vary between different platforms.

Therefore, the objective of the study is to characterize the pattern of radiolabeled tracer uptake in noninfected transcatheter heart valves in early follow-up after TAVR.

This will be a pilot study including 30 patients after TAVR procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18-year-old undergoing TAVR procedure with Edwards Sapien 3 and Core Valve Evolut R devices.
* Informed written consent

Exclusion Criteria:

* Inability to provide signed informed consent.
* Patients with definitive or possible IE according to modified Duke criteria and current clinical guidelines for the management of IE.
* Any contraindication for 18F-FDG PET/CT.
* Any condition making it unlikely the patient will be able to complete the protocol procedures and follow-up visits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing TAVR procedure with Edwards Sapien 3 and Core Valve Evolut R devices.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-11-09 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Radiolabeled tracer uptake grade (intense, moderate, mild or absent) in the prosthetic and periprosthetic areas. | 3 months after TAVR
  Visual analysis grading the radiolabeled tracer molecules uptake in the prosthetic and periprosthetic areas as intense, moderate, mild or absent. This visual analysis will be defined whether the PET/CT was positive (intense/moderate) or negative (mild/absent).

SECONDARY OUTCOMES:
Maximal standardized uptake value (SUVmax) using an average of 3 measurements from 3 volumes of interest (5mm3) introduced in the prosthetic region at equal distances from each other. | 3 months after TAVR
  The intensity of the radiolabeled tracer uptake will be determined by measuring the maximal standardized uptake value (SUVmax)), which is obtained by normalizing the tissue concentration of the radiolabeled tracer activity and the patient's weight. SUVmax will be calculated using an average of 3 measurements from 3 volumes of interest (5mm3) introduced in the prosthetic region at equal distances from each other. The prosthetic valve-to-background ratio will be calculated by dividing the prosthetic valve SUV max by the atrial blood SUVmax.
Differences in radiolabeled tracer uptake grade in the prosthetic and periprosthetic areas between the Edwards valve versus the CoreValve valve. | 3 months after TAVR
  Differences in radiolabeled tracer uptake pattern with different valves: Edwards THV vs CoreValve THV
Correlation between radiolabeled tracer uptake grade and time from TAVR | 3 months after TAVR
  Relationship between radiolabeled tracer uptake and time from the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche de L'Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vongpatanasin W, Hillis LD, Lange RA. Prosthetic heart valves. N Engl J Med. 1996 Aug 8;335(6):407-16. doi: 10.1056/NEJM199608083350607. No abstract available. PMID 8676934
- [Background] Hoen B, Duval X. Clinical practice. Infective endocarditis. N Engl J Med. 2013 Apr 11;368(15):1425-33. doi: 10.1056/NEJMcp1206782. No abstract available. PMID 23574121
- [Background] Wang A, Pappas P, Anstrom KJ, Abrutyn E, Fowler VG Jr, Hoen B, Miro JM, Corey GR, Olaison L, Stafford JA, Mestres CA, Cabell CH; International Collaboration on Endocarditis Investigators. The use and effect of surgical therapy for prosthetic valve infective endocarditis: a propensity analysis of a multicenter, international cohort. Am Heart J. 2005 Nov;150(5):1086-91. doi: 10.1016/j.ahj.2005.01.023. PMID 16291003
- [Background] Akowuah EF, Davies W, Oliver S, Stephens J, Riaz I, Zadik P, Cooper G. Prosthetic valve endocarditis: early and late outcome following medical or surgical treatment. Heart. 2003 Mar;89(3):269-72. doi: 10.1136/heart.89.3.269. PMID 12591827
- [Background] Edwards MB, Ratnatunga CP, Dore CJ, Taylor KM. Thirty-day mortality and long-term survival following surgery for prosthetic endocarditis: a study from the UK heart valve registry. Eur J Cardiothorac Surg. 1998 Aug;14(2):156-64. doi: 10.1016/s1010-7940(98)00148-1. PMID 9755001
- [Background] Tornos P, Almirante B, Olona M, Permanyer G, Gonzalez T, Carballo J, Pahissa A, Soler-Soler J. Clinical outcome and long-term prognosis of late prosthetic valve endocarditis: a 20-year experience. Clin Infect Dis. 1997 Mar;24(3):381-6. doi: 10.1093/clinids/24.3.381. PMID 9114189
- [Background] Grover FL, Cohen DJ, Oprian C, Henderson WG, Sethi G, Hammermeister KE. Determinants of the occurrence of and survival from prosthetic valve endocarditis. Experience of the Veterans Affairs Cooperative Study on Valvular Heart Disease. J Thorac Cardiovasc Surg. 1994 Aug;108(2):207-14. PMID 8041168
- [Background] Smith CR, Leon MB, Mack MJ, Miller DC, Moses JW, Svensson LG, Tuzcu EM, Webb JG, Fontana GP, Makkar RR, Williams M, Dewey T, Kapadia S, Babaliaros V, Thourani VH, Corso P, Pichard AD, Bavaria JE, Herrmann HC, Akin JJ, Anderson WN, Wang D, Pocock SJ; PARTNER Trial Investigators. Transcatheter versus surgical aortic-valve replacement in high-risk patients. N Engl J Med. 2011 Jun 9;364(23):2187-98. doi: 10.1056/NEJMoa1103510. Epub 2011 Jun 5. PMID 21639811
- [Background] Adams DH, Popma JJ, Reardon MJ, Yakubov SJ, Coselli JS, Deeb GM, Gleason TG, Buchbinder M, Hermiller J Jr, Kleiman NS, Chetcuti S, Heiser J, Merhi W, Zorn G, Tadros P, Robinson N, Petrossian G, Hughes GC, Harrison JK, Conte J, Maini B, Mumtaz M, Chenoweth S, Oh JK; U.S. CoreValve Clinical Investigators. Transcatheter aortic-valve replacement with a self-expanding prosthesis. N Engl J Med. 2014 May 8;370(19):1790-8. doi: 10.1056/NEJMoa1400590. Epub 2014 Mar 29. PMID 24678937
- [Background] Leon MB, Smith CR, Mack MJ, Makkar RR, Svensson LG, Kodali SK, Thourani VH, Tuzcu EM, Miller DC, Herrmann HC, Doshi D, Cohen DJ, Pichard AD, Kapadia S, Dewey T, Babaliaros V, Szeto WY, Williams MR, Kereiakes D, Zajarias A, Greason KL, Whisenant BK, Hodson RW, Moses JW, Trento A, Brown DL, Fearon WF, Pibarot P, Hahn RT, Jaber WA, Anderson WN, Alu MC, Webb JG; PARTNER 2 Investigators. Transcatheter or Surgical Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2016 Apr 28;374(17):1609-20. doi: 10.1056/NEJMoa1514616. Epub 2016 Apr 2. PMID 27040324
- [Background] Reardon MJ, Van Mieghem NM, Popma JJ, Kleiman NS, Sondergaard L, Mumtaz M, Adams DH, Deeb GM, Maini B, Gada H, Chetcuti S, Gleason T, Heiser J, Lange R, Merhi W, Oh JK, Olsen PS, Piazza N, Williams M, Windecker S, Yakubov SJ, Grube E, Makkar R, Lee JS, Conte J, Vang E, Nguyen H, Chang Y, Mugglin AS, Serruys PW, Kappetein AP; SURTAVI Investigators. Surgical or Transcatheter Aortic-Valve Replacement in Intermediate-Risk Patients. N Engl J Med. 2017 Apr 6;376(14):1321-1331. doi: 10.1056/NEJMoa1700456. Epub 2017 Mar 17. PMID 28304219
- [Background] Baumgartner H, Falk V, Bax JJ, De Bonis M, Hamm C, Holm PJ, Iung B, Lancellotti P, Lansac E, Rodriguez Munoz D, Rosenhek R, Sjogren J, Tornos Mas P, Vahanian A, Walther T, Wendler O, Windecker S, Zamorano JL; ESC Scientific Document Group. 2017 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2017 Sep 21;38(36):2739-2791. doi: 10.1093/eurheartj/ehx391. No abstract available. PMID 28886619
- [Background] Regueiro A, Linke A, Latib A, Ihlemann N, Urena M, Walther T, Husser O, Herrmann HC, Nombela-Franco L, Cheema AN, Le Breton H, Stortecky S, Kapadia S, Bartorelli AL, Sinning JM, Amat-Santos I, Munoz-Garcia A, Lerakis S, Gutierrez-Ibanes E, Abdel-Wahab M, Tchetche D, Testa L, Eltchaninoff H, Livi U, Castillo JC, Jilaihawi H, Webb JG, Barbanti M, Kodali S, de Brito FS Jr, Ribeiro HB, Miceli A, Fiorina C, Dato GM, Rosato F, Serra V, Masson JB, Wijeysundera HC, Mangione JA, Ferreira MC, Lima VC, Carvalho LA, Abizaid A, Marino MA, Esteves V, Andrea JC, Giannini F, Messika-Zeitoun D, Himbert D, Kim WK, Pellegrini C, Auffret V, Nietlispach F, Pilgrim T, Durand E, Lisko J, Makkar RR, Lemos PA, Leon MB, Puri R, San Roman A, Vahanian A, Sondergaard L, Mangner N, Rodes-Cabau J. Association Between Transcatheter Aortic Valve Replacement and Subsequent Infective Endocarditis and In-Hospital Death. JAMA. 2016 Sep 13;316(10):1083-92. doi: 10.1001/jama.2016.12347. PMID 27623462
- [Background] Habib G, Lancellotti P, Antunes MJ, Bongiorni MG, Casalta JP, Del Zotti F, Dulgheru R, El Khoury G, Erba PA, Iung B, Miro JM, Mulder BJ, Plonska-Gosciniak E, Price S, Roos-Hesselink J, Snygg-Martin U, Thuny F, Tornos Mas P, Vilacosta I, Zamorano JL; ESC Scientific Document Group. 2015 ESC Guidelines for the management of infective endocarditis: The Task Force for the Management of Infective Endocarditis of the European Society of Cardiology (ESC). Endorsed by: European Association for Cardio-Thoracic Surgery (EACTS), the European Association of Nuclear Medicine (EANM). Eur Heart J. 2015 Nov 21;36(44):3075-3128. doi: 10.1093/eurheartj/ehv319. Epub 2015 Aug 29. No abstract available. PMID 26320109
- [Background] Gomes A, Glaudemans AWJM, Touw DJ, van Melle JP, Willems TP, Maass AH, Natour E, Prakken NHJ, Borra RJH, van Geel PP, Slart RHJA, van Assen S, Sinha B. Diagnostic value of imaging in infective endocarditis: a systematic review. Lancet Infect Dis. 2017 Jan;17(1):e1-e14. doi: 10.1016/S1473-3099(16)30141-4. Epub 2016 Oct 18. PMID 27746163
- [Background] Mathieu C, Mikail N, Benali K, Iung B, Duval X, Nataf P, Jondeau G, Hyafil F, Le Guludec D, Rouzet F. Characterization of 18F-Fluorodeoxyglucose Uptake Pattern in Noninfected Prosthetic Heart Valves. Circ Cardiovasc Imaging. 2017 Mar;10(3):e005585. doi: 10.1161/CIRCIMAGING.116.005585. PMID 28298285
- [Background] Sarrazin JF, Philippon F, Trottier M, Tessier M. Role of radionuclide imaging for diagnosis of device and prosthetic valve infections. World J Cardiol. 2016 Sep 26;8(9):534-546. doi: 10.4330/wjc.v8.i9.534. PMID 27721936